CLINICAL TRIAL: NCT04413851
Title: A Feasibility Study to Evaluate Passive Collection of Activity Data in Subjects With Agitation in the Context of Dementia
Brief Title: Feasibility of Passive Data Collection in Dementia Subjects With Agitation
Status: Completed | Type: Observational
Sponsor: HealthMode Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HM060401
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Dementia; Alzheimer Disease; Vascular Dementia; Frontotemporal Dementia; Lewy Body Dementia; Mixed Dementia
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Frontotemporal Dementia; Lewy Body Disease; Mixed Dementias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dementia: Subjects with a diagnosis of dementia who are experiencing agitation severe enough that it interferes with activities of daily living or social interaction.

SUMMARY:
This is a multi-center, observational, feasibility study, to evaluate long term passive data collection, data quality, and user experience of HealthMode Agitation (Apps) to collect motion, location, physiological, and audio data; and eCOA and EMA responses with mobile devices (iPhone, Apple Watch).

The purpose of this study is to evaluate and improve HealthMode Apps data collection and usability in subjects experiencing agitation in the context of dementia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years and older.
* Subjects who have met DSM-5 criteria for Dementia (all cause)
* Subjects with a recent history of agitation in the past 6 months to a point that impairs social activities, requires staffing or medical intervention (kick, bite, flailing, etc.), impairs ability for functional activities of daily living, as disclosed by a caregiver or documented in the medical record.
* Subjects resident in a group home, nursing home, or assisted living are eligible to participate.
* Subjects who can read, understand and provide written informed consent or who have a Legally Acceptable Representative (LAR)
* Subjects who are willing and able to carry a smartphone and wear an activity tracker on their wrist or hand, alone or with the help of a caregiver.
* Subjects who, either alone or with a caregiver, are able to operate a smartphone and wrist or hand-worn activity tracker, alone or with the help of a caregiver.
* Subjects who are in good general health prior to study participation as determined by a detailed medical history, and in the opinion of the Principal Investigator.
* Subjects, who are able to ambulate without an assistive device, or with a single point cane.

Exclusion Criteria:

* Subjects who are unwilling or unable to carry a smartphone and wear an activity tracker on their wrist or hand.
* Subjects with serious or unstable medical illnesses. These include current hepatic (moderate-severe hepatic impairment), renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease, congestive heart failure), endocrinologic, neurologic or hematologic disease.
* Subjects who are considered by the investigator, for any reason, to be an unsuitable candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible individuals who have a diagnosis of dementia and a recent history of agitation will sign an informed consent, with a legally authorized representative (LAR) when necessary, to enroll in the study.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of passive and continuous data collection | 28 days
  Total time and percentage of continuous data collection for each stream of data aiming for >50% coverage.

SECONDARY OUTCOMES:
Tolerability of carrying a smartphone and wearing a data collection sensor on the wrist and/or hand in a population of subjects who may have frequent episodes of agitation or impulsive behavior. | 28 days
  Caregiver and Staff engagement with the eCOA and EMA (threshold 80% completion) and responses to usability questionnaires at week 1 and 4 to provide feedback on comfort, usability and engagement. The score ranges from 10 to 50, higher score indicating a better usability.

OTHER OUTCOMES:
Suitability of individual data streams and their combinations for purposes of identification of agitation episodes in passively collected data. | 28 days
  Comparison of data collected from the smartphone and wearable device to episodes identified by subject or caregiver assessment:
  1. Cleaned single channel data compared to assessments
  2. Cleaned multichannel data compared to assessments
  3. Analyzed multichannel data compared to assessments
  4. Subject/Caregiver assessment data compared to agitation scale ratings
  5. Agitation scale ratings compared to cleaned single and multichannel data and analyzed multichannel data.
  6. Merged subject/caregiver assessment and multichannel data compared to agitation scale ratings

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tucson Neuroscience Research, LLC, Tucson, Arizona
  - Virtual Research Site, New York, New York